CLINICAL TRIAL: NCT00590512
Title: Dietary Salt Intake and Vascular Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rhonda Bentley-Lewis, MD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2004P002705
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: dietary salt; sodium; blood vessels; vascular function; endothelial function; heart disease risk; cardiovascular disease risk
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Sodium (Active Comparator): High sodium
  Interventions: Dietary Supplement: High sodium
- Low sodium (Active Comparator): Low sodium
  Interventions: Dietary Supplement: Low sodium

INTERVENTIONS:
Dietary Supplement: High sodium
  Arms: High Sodium
Dietary Supplement: Low sodium
  Arms: Low sodium

SUMMARY:
The purpose of this study is to look at the effects of high- and low-salt diets on blood vessel function in healthy subjects.

DETAILED DESCRIPTION:
Healthy volunteers will be enrolled in a dietary sodium intervention to examine impact on vascular function.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, African-American volunteers
2. 18-35 years of age,
3. No personal or first degree relative with hypertension or diabetes,
4. Blood pressure <130/85 mmHg and > 90/60 at the screening visit,
5. Body mass index <30 kg/m2,
6. No clinically significant abnormalities on screening tests (complete blood count, serum electrolytes, liver enzymes, thyroid stimulating hormone, urinalysis and electrocardiogram).

Exclusion Criteria:

1. Alcohol intake >2 beverage/night,
2. Smoking,
3. Recreational drug use,
4. Personal history of coronary disease, diabetes, hypertension, stroke, kidney disease, or illness requiring overnight hospitalization in the past 6 months,
5. Prescription or herbal medication use,
6. Ischemic changes on resting electrocardiogram,
7. Known hypersensitivity to any of the study drugs,
8. Other active medical problems detected by examination or laboratory testing.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2005-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
endothelial function | one week

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Bentley-Lewis, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States